CLINICAL TRIAL: NCT01266993
Title: Persistence of Antibodies After Vaccination With a Dose of GSK Biologicals' Meningococcal Vaccine GSK134612 in Healthy Children and Safety and Immunogenicity of a Booster Dose at 68 Months Post-primary Vaccination
Brief Title: Persistence and Booster Study of GSK Biologicals' Meningococcal Vaccine (GSK134612) in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113977; 2010-018730-51 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-24 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Infections, Meningococcal; Meningococcal Vaccines
Keywords: Immunogenicity; Persistence; Safety; Conjugate vaccine; Meningococcal vaccine
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimenrix Group (Experimental): Healthy male or female subjects aged 2 through 10 years old, who were primed with one dose of Nimenrix vaccine during the primary 111414 study (NCT00674583), additionally received one booster dose of Nimenrix vaccine in the current study, at Month 68, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Nimenrix (GSK134612 vaccine)
- Menjugate Group (Experimental): Healthy male or female subjects aged 2 through 10 years old, who were primed with one dose of Menjugate vaccine during the primary 111414 study (NCT00674583), additionally received one booster dose of Menjugate vaccine in the current study, at Month 68, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Menjugate

INTERVENTIONS:
Biological: Nimenrix (GSK134612 vaccine) — Intramuscular, 1 dose
  Arms: Nimenrix Group
Biological: Menjugate — Intramuscular, 1 dose
  Arms: Menjugate Group

SUMMARY:
The purpose of the study is to evaluate the persistence of the immune response of GSK134612 vaccine up to 68 months after vaccination in the primary vaccination study (NCT number = NCT00674583) of 2 to 10 year old subjects. This study will also evaluate the safety and immunogenicity of a booster dose of GSK134612 vaccine subjects who were primed in the primary vaccination study with either GSK134612 vaccine or Menjugate®.

This protocol posting deals with objectives & outcome measures of the persistence and booster epochs. The objectives & outcome measures of the primary epoch are presented in a separate protocol posting (NCT number = NCT00674583)

DETAILED DESCRIPTION:
Subjects were previously vaccinated at 2 to 10 years of age with GSK134612 or with Menjugate®. The persistence phase starts 32 months after the primary vaccination and blood samples will be taken at 32, 44, 56 and 68 months after primary vaccination. All subjects will receive a booster dose of GSK134612 at 68 months after primary vaccination and a blood sample will be taken 1 month after administration of the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female who was primed with MenACWY-TT or Menjugate in the primary vaccination study (NCT number = NCT00674583).
* Written informed consent obtained from the parent(s)/Legally Acceptable Representatives(s) of the subject and written informed assent obtained from the subject (at investigator discretion).
* Healthy subjects as established by medical history and clinical examination before entering into the study.

All subjects must meet the additional following criteria prior to receiving the booster vaccination:

* Subjects who had a blood sample taken at Visit 4 during the persistence epoch of the current study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product within 30 days preceding the first persistence blood sample or planned use within 30 days preceding a blood sample during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs during the study period. (For corticosteroids, prednisone <10 mg/day, or equivalent, inhaled and topical steroids are allowed).
* Concurrently participating in another clinical study or planned participation in another clinical study, in which the subject has been or will be exposed to an investigational or a non-investigational product within 30 days of a blood sample.
* History of meningococcal disease.
* Administration of a meningococcal polysaccharide or a meningococcal polysaccharide conjugate vaccine since the previous vaccination in the primary vaccination study (NCT number = NCT00674583).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection, based on medical history and physical examination.
* Serious chronic illness.
* Administration of immunoglobulins and/or blood products within the 3 months preceding the subject's first visit.
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* Subjects in contact with somebody suffering from an invasive infection with meningococcal serogroups A, C, Y or W-135.
* Subjects living in a geographic area where local outbreak with meningococcal serogroup C has occurred.

Exclusion criteria for booster vaccination to be checked at Visit 4 (Month 68)

* Child in care.
* Use of any investigational or non-registered product within 30 days preceding the booster vaccination or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccination. (For corticosteroids, prednisone <10 mg/day, or equivalent, inhaled and topical steroids are allowed).
* Vaccination with meningococcal polysaccharide or conjugate vaccine of serogroup A, B, C, W-135, and/or Y since the previous vaccination in the primary vaccination study (NCT number = NCT00674583).
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection, based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster vaccination or planned administration during the study period.
* Concurrently participating in another clinical study or planned participation in another clinical study, at any time during the study period, (from the time of the booster until the end of the study) in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* Hypersensitivity to latex.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within the last 30 days of the dose of vaccine(s) with the exception of a licensed inactivated influenza vaccine.
* Previous vaccination with tetanus toxoids within the last 30 days.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Serious chronic illness.
* History of any neurological disorders or seizures (although subjects with a prior history of a single episode of benign febrile seizures may be allowed to participate in the study).
* Acute disease and/or fever at the time of vaccination.
* History of chronic alcohol consumption and/or drug abuse.
* History of hypotonic-hyporesponsive episodes (HHEs) following vaccination.
* Subjects in contact with somebody suffering from an invasive infection with meningococcal serogroups A, C, Y or W-135.
* Subjects living in a geographic area where local outbreak with meningococcal serogroup C has occurred.
* Pregnant or lactating female.
* Female of child-bearing potential planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 271 (Actual)
Dates: Start 2011-01-03 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- France (8):
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Lingolsheim
  - GSK Investigational Site, Miribel
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Laurent-du-Var
  - GSK Investigational Site, Tours
- Germany (12):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Berlin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 282 subjects participating to the study, 271 participated to Month 32-44 period, 261 to Month 44-56, 260 to Month 56-68, and 282 to Month 68-69 booster period.
  Out of 282 subjects participating to Month 68-69 booster period, 41 subjects had a subject number allocated but received no vaccine dose, hence only 241 started this phase.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Menjugate Group: Healthy male or female subjects aged 2 through 10 years old, who were primed with one dose of Menjugate vaccine during the primary 111414 study (NCT00674583), additionally received one booster dose of Nimenrix vaccine in the current study, at Month 68, administered intramuscularly in the deltoid region of the non-dominant arm.
Period: Persistence Phase (Month 32-44)
Arm/Group | Nimenrix Group | Menjugate Group
Started | 199 | 72
Completed | 199 | 72
Not Completed | 0 | 0
Period: Persistence Phase (Month 44-56)
Arm/Group | Nimenrix Group | Menjugate Group
Started | 193 | 68
Completed | 193 | 68
Not Completed | 0 | 0
Period: Persistence Phase (Month 56-68)
Arm/Group | Nimenrix Group | Menjugate Group
Started | 193 | 67
Completed | 193 | 67
Not Completed | 0 | 0
Period: Booster Phase (Month 68-69)
Arm/Group | Nimenrix Group | Menjugate Group
Started | 179 | 62
Completed | 174 | 60
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix Group | Menjugate Group | Total
Number analyzed (Participants) | 199 | 72 | 271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.4 (2.58) | 8.1 (2.42) | 8.32 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 34 | 137
  Male | 96 | 38 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage / African American | 7 | 2 | 9
  Geographic ancestry: American Indian or Alaskan native | 0 | 0 | 0
  Geographic ancestry: Asian - Central/South Asian heritage | 1 | 0 | 1
  Geographic ancestry: Asian - East Asian heritage | 1 | 1 | 2
  Geographic ancestry: Asian - Japanese heritage | 0 | 0 | 0
  Geographic ancestry: Asian - South East Asian heritage | 1 | 0 | 1
  Geographic ancestry: Native Hawaiian or other pacific islander | 0 | 0 | 0
  Geographic ancestry: White - Arabic / North African heritage | 12 | 6 | 18
  Geographic ancestry: White - Caucasian/European Heritage | 169 | 61 | 230
  Geographic ancestry: Other | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay, Using Baby Rabbit Complement, Against Neisseria Meningitides Serogroup A, C, W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) Antibody Titers Was Greater Than or Equal to (≥) 1:8, at Month 32.
Description: The pre-defined cut-off value of the assay for the rSBA titers was greater than or equal to (≥) 1:8. These analyses have been performed by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 32, post-primary vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for persistence at Month 32, which included all evaluable subjects primed during the primary 111414 study (NCT00674583) according to their treatment group, for whom assay results were available for at least one tested antigen at Month 32.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 193 | 69
Participants
  rSBA-MenA | 167 | 15
  rSBA-MenC: number analyzed (Participants) | 192 | 69
  rSBA-MenC | 124 | 53
  rSBA-MenW-135 | 149 | 5
  rSBA-MenY | 157 | 10

2. Primary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:8, at Month 44.
Description: as for outcome 1
Time Frame: At Month 44, post-primary vaccination
Population: The analysis was performed on the ATP cohort for persistence at Month 44, which included all evaluable subjects primed during the primary 111414 study (NCT00674583) according to their treatment group, for whom assay results were available for at least one tested antigen at Month 44.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 189 | 66
Participants
  rSBA-MenA | 162 | 17
  rSBA-MenC | 70 | 30
  rSBA-MenW-135 | 129 | 7
  rSBA-MenY | 118 | 4

3. Primary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:8, at Month 56.
Description: as for outcome 1
Time Frame: At Month 56, post-primary vaccination
Population: The analysis was performed on the ATP cohort for persistence at Month 56, which included all evaluable subjects primed during the primary 111414 study (NCT00674583) according to their treatment group, for whom assay results were available for at least one tested antigen at Month 56.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 186 | 65
Participants
  rSBA-MenA | 161 | 19
  rSBA-MenC | 110 | 42
  rSBA-MenW-135 | 145 | 17
  rSBA-MenY: number analyzed (Participants) | 186 | 64
  rSBA-MenY | 149 | 14

4. Primary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:8, at Month 68.
Description: as for outcome 1
Time Frame: At Month 68, post-primary vaccination
Population: The analysis was performed on the ATP cohort for persistence at Month 68, which included all evaluable subjects primed during the primary 111414 study (NCT00674583) according to their treatment group, for whom assay results were available for at least one tested antigen at Month 68.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 178 | 61
Participants
  rSBA-MenA | 154 | 18
  rSBA-MenC | 71 | 38
  rSBA-MenW-135 | 94 | 9
  rSBA-MenY | 127 | 8

5. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:128, at Month 32.
Description: The pre-defined cut-off value of the assay for the rSBA titers was greater than or equal to (≥) 1:128. These analyses have been performed by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 32, post-primary vaccination
Population: The analysis was performed on the ATP cohort for persistence at Month 32, which included all evaluable subjects primed during the primary 111414 study (NCT00674583) according to their treatment group, for whom assay results were available for at least one tested antigen at Month 32.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 193 | 69
Participants
  rSBA-MenA | 140 | 9
  rSBA-MenC: number analyzed (Participants) | 192 | 69
  rSBA-MenC | 69 | 35
  rSBA-MenW-135 | 136 | 5
  rSBA-MenY | 145 | 8

6. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:128, at Month 44.
Description: as for outcome 5
Time Frame: At Month 44, post-primary vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 189 | 66
Participants
  rSBA-MenA | 151 | 16
  rSBA-MenC | 38 | 23
  rSBA-MenW-135 | 120 | 5
  rSBA-MenY | 107 | 3

7. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:128, at Month 56.
Description: as for outcome 5
Time Frame: At Month 56, post-primary vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 186 | 65
Participants
  rSBA-MenA | 107 | 10
  rSBA-MenC | 65 | 32
  rSBA-MenW-135 | 123 | 10
  rSBA-MenY: number analyzed (Participants) | 186 | 64
  rSBA-MenY | 139 | 10

8. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:128, at Month 68.
Description: as for outcome 5
Time Frame: At Month 68, post-primary vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 178 | 61
Participants
  rSBA-MenA | 107 | 12
  rSBA-MenC | 38 | 25
  rSBA-MenW-135 | 84 | 8
  rSBA-MenY | 118 | 6

9. Secondary Outcome: Antibody Titers for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY, at Month 32.
Description: Antibody titers were presented as geometric mean titers (GMTs). These analyses were performed by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 32, post-primary vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 193 | 69
Titers
  rSBA-MenA | 196.3 [144.1 to 267.2] | 8 [5.5 to 11.7]
  rSBA-MenC: number analyzed (Participants) | 192 | 69
  rSBA-MenC | 34.8 [26 to 46.4] | 86.5 [47.3 to 158.1]
  rSBA-MenW-135 | 213.9 [149.3 to 306.6] | 5.6 [4.2 to 7.6]
  rSBA-MenY | 227.4 [164.8 to 313.7] | 7.2 [5 to 10.4]

10. Secondary Outcome: Antibody Titers for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY, at Month 44.
Description: as for outcome 9
Time Frame: At Month 44, post-primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 189 | 66
Titers
  rSBA-MenA | 307.5 [223.7 to 422.8] | 13.5 [8 to 23]
  rSBA-MenC | 14.5 [10.9 to 19.2] | 31 [16.6 to 58]
  rSBA-MenW-135 | 103.5 [72.5 to 147.6] | 5.9 [4.3 to 8.1]
  rSBA-MenY | 78.9 [54.6 to 114] | 4.9 [3.9 to 6.2]

11. Secondary Outcome: Antibody Titers for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY, at Month 56.
Description: as for outcome 9
Time Frame: At Month 56, post-primary vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 186 | 65
Titers
  rSBA-MenA | 120.1 [87.0 to 165.9] | 9.8 [6.4 to 15.0]
  rSBA-MenC | 30.5 [22.6 to 41.1] | 69.0 [36.9 to 128.9]
  rSBA-MenW-135 | 158.3 [112.4 to 222.9] | 10.3 [6.4 to 16.6]
  rSBA-MenY: number analyzed (Participants) | 186 | 64
  rSBA-MenY | 233.2 [166.0 to 327.6] | 9.0 [6.0 to 13.6]

12. Secondary Outcome: Antibody Titers for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY, at Month 68.
Description: as for outcome 9
Time Frame: At Month 68, post-primary vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 178 | 61
Titers
  rSBA-MenA | 129.5 [93.5 to 179.3] | 11.1 [7.0 to 17.7]
  rSBA-MenC | 14.2 [10.8 to 18.7] | 44.5 [23.7 to 83.6]
  rSBA-MenW-135 | 59.2 [39.3 to 89.2] | 7.8 [5.0 to 12.1]
  rSBA-MenY | 139.4 [96.0 to 202.5] | 6.8 [4.6 to 10.2]

13. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay, Using Human Complement, Against N. Meningitides Serogroup A, C, W-135, Y (hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY) Antibody Titers ≥ 1:4 and ≥ 1:8, at Month 32.
Description: The pre-defined cut-off values of the assay for the hSBA titers were greater than or equal to (≥) 1:4 and ≥ 1:8. These analyses have been performed on 50% of the subjects in each group, by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 32, post-primary vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 91 | 34
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 90 | 34
  hSBA-MenA, ≥ 1:4 | 24 | 5
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 90 | 33
  hSBA-MenC, ≥ 1:4 | 86 | 30
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 86 | 23
  hSBA-MenW-135, ≥ 1:4 | 73 | 4
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 91 | 28
  hSBA-MenY, ≥ 1:4 | 74 | 13
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 90 | 34
  hSBA-MenA, ≥ 1:8 | 23 | 5
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 90 | 33
  hSBA-MenC, ≥ 1:8 | 86 | 30
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 86 | 23
  hSBA-MenW-135, ≥ 1:8 | 73 | 4
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 91 | 28
  hSBA-MenY, ≥ 1:8 | 74 | 13

14. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers ≥ 1:4 and ≥ 1:8, at Month 44.
Description: as for outcome 13
Time Frame: At Month 44, post-primary vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 89 | 31
Participants
  hSBA-MenA, ≥ 1:4 | 26 | 5
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 82 | 31
  hSBA-MenC, ≥ 1:4 | 63 | 20
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 87 | 30
  hSBA-MenW-135, ≥ 1:4 | 70 | 8
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 76 | 26
  hSBA-MenY, ≥ 1:4 | 63 | 12
  hSBA-MenA, ≥ 1:8 | 23 | 5
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 82 | 31
  hSBA-MenC, ≥ 1:8 | 63 | 20
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 87 | 30
  hSBA-MenW-135, ≥ 1:8 | 70 | 8
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 76 | 26
  hSBA-MenY, ≥ 1:8 | 63 | 12

15. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers ≥ 1:4 and ≥ 1:8, at Month 56.
Description: as for outcome 13
Time Frame: At Month 56, post-primary vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 89 | 33
Participants
  hSBA-MenA, ≥ 1:4 | 53 | 19
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 86 | 31
  hSBA-MenC, ≥ 1:4 | 66 | 21
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 83 | 30
  hSBA-MenW-135, ≥ 1:4 | 69 | 13
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 89 | 31
  hSBA-MenY, ≥ 1:4 | 79 | 22
  hSBA-MenA, ≥ 1:8 | 53 | 19
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 86 | 31
  hSBA-MenC, ≥ 1:8 | 64 | 21
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 83 | 30
  hSBA-MenW-135, ≥ 1:8 | 69 | 13
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 89 | 31
  hSBA-MenY, ≥ 1:8 | 79 | 22

16. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers ≥ 1:4 and ≥ 1:8, at Month 68.
Description: The pre-defined cut-off values of the assay for the hSBA titers were greater than or equal to (≥) 1:4 and ≥ 1:8. These analyses have been performed in all subjects, by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 68, post-primary vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 172 | 59
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 170 | 59
  hSBA-MenA, ≥ 1:4 | 70 | 23
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 172 | 57
  hSBA-MenC, ≥ 1:4 | 134 | 43
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 159 | 52
  hSBA-MenW-135, ≥ 1:4 | 125 | 19
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 159 | 58
  hSBA-MenY, ≥ 1:4 | 116 | 24
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 170 | 59
  hSBA-MenA, ≥ 1:8 | 69 | 21
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 172 | 57
  hSBA-MenC, ≥ 1:8 | 130 | 43
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 159 | 52
  hSBA-MenW-135, ≥ 1:8 | 125 | 19
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 159 | 58
  hSBA-MenY, ≥ 1:8 | 116 | 24

17. Secondary Outcome: Antibody Titers for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY, at Month 32.
Description: Antibody titers were presented as geometric mean titers (GMTs). These analyses were performed on 50% of the subjects in each group, by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 32, post-primary vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 91 | 34
Titers
  hSBA-MenA: number analyzed (Participants) | 90 | 34
  hSBA-MenA | 4.6 [3.3 to 6.3] | 2.7 [2.1 to 3.4]
  hSBA-MenC: number analyzed (Participants) | 90 | 33
  hSBA-MenC | 75.9 [53.4 to 107.9] | 82.2 [34.6 to 195.8]
  hSBA-MenW-135: number analyzed (Participants) | 86 | 23
  hSBA-MenW-135 | 69.9 [48.2 to 101.5] | 3.8 [2 to 7.1]
  hSBA-MenY: number analyzed (Participants) | 91 | 28
  hSBA-MenY | 79.2 [52.5 to 119.3] | 15.1 [6.3 to 36.5]

18. Secondary Outcome: Antibody Titers for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY, at Month 44.
Description: as for outcome 17
Time Frame: At Month 44, post-primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 89 | 31
Titers
  hSBA-MenA | 4.8 [3.4 to 6.7] | 2.8 [2.1 to 3.7]
  hSBA-MenC: number analyzed (Participants) | 82 | 31
  hSBA-MenC | 36.4 [23.1 to 57.2] | 38.8 [13.3 to 113.2]
  hSBA-MenW-135: number analyzed (Participants) | 87 | 30
  hSBA-MenW-135 | 64.3 [42.7 to 96.8] | 5.2 [2.8 to 9.5]
  hSBA-MenY: number analyzed (Participants) | 76 | 26
  hSBA-MenY | 126.7 [78 to 205.7] | 16.8 [16.8 to 44.9]

19. Secondary Outcome: Antibody Titers for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY, at Month 56.
Description: as for outcome 17
Time Frame: At Month 56, post-primary vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 89 | 33
Titers
  hSBA-MenA | 10.6 [7.6 to 14.9] | 7.6 [5.0 to 11.8]
  hSBA-MenC: number analyzed (Participants) | 86 | 31
  hSBA-MenC | 20.6 [13.8 to 30.8] | 31.2 [11.5 to 85.0]
  hSBA-MenW-135: number analyzed (Participants) | 83 | 30
  hSBA-MenW-135 | 59.3 [40.2 to 87.6] | 9.2 [4.7 to 18.2]
  hSBA-MenY: number analyzed (Participants) | 89 | 31
  hSBA-MenY | 117.9 [80.8 to 171.9] | 35.7 [16.8 to 75.9]

20. Secondary Outcome: Antibody Titers for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY, at Month 68.
Description: as for outcome 9
Time Frame: At Month 68, post-primary vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 172 | 59
Titers
  hSBA-MenA: number analyzed (Participants) | 170 | 59
  hSBA-MenA | 6.9 [5.4 to 8.9] | 4.5 [3.3 to 6.0]
  hSBA-MenC: number analyzed (Participants) | 172 | 57
  hSBA-MenC | 28.4 [21.2 to 37.9] | 34.3 [19.0 to 61.0]
  hSBA-MenW-135: number analyzed (Participants) | 159 | 52
  hSBA-MenW-135 | 56.7 [41.5 to 77.3] | 8.1 [4.7 to 13.8]
  hSBA-MenY: number analyzed (Participants) | 159 | 58
  hSBA-MenY | 56.3 [39.5 to 80.3] | 13.3 [7.0 to 25.1]

21. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ 1:128 and 1:8.
Description: The pre-defined cut-off values of the assay for the rSBA titers were greater than or equal to (≥) 1:128 and ≥ 1:8. These analyses have been performed by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 69, one month post-booster vaccination
Population: The analysis was performed on the Booster ATP cohort for immunogenicity, which included all evaluable subjects from the Booster ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after the booster vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 165 | 55
Participants
  rSBA-MenA, ≥ 1:8 | 165 | 55
  rSBA-MenC, ≥ 1:8 | 165 | 55
  rSBA-MenW-135, ≥ 1:8 | 165 | 55
  rSBA-MenY, ≥ 1:8 | 165 | 55
  rSBA-MenA, ≥ 1:128 | 165 | 55
  rSBA-MenC, ≥ 1:128 | 165 | 55
  rSBA-MenW-135, ≥ 1:128 | 165 | 55
  rSBA-MenY, ≥ 1:128 | 165 | 55

22. Secondary Outcome: Antibody Titers for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY
Description: as for outcome 9
Time Frame: At Month 69, one month post-booster vaccination
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 165 | 55
Titers
  rSBA-MenA | 5613.0 [4946.3 to 6369.4] | 3521.1 [2912.5 to 4256.9]
  rSBA-MenC | 5314.6 [4596.2 to 6145.4] | 7042.2 [5317.4 to 9326.5]
  rSBA-MenW-135 | 14750.6 [12779.6 to 17025.6] | 10540.4 [8455.2 to 13139.8]
  rSBA-MenY | 7954.6 [7167.8 to 8827.8] | 5829.2 [4725.6 to 7190.6]

23. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers ≥ 1:4 and 1:8.
Description: The pre-defined cut-off values of the assay for the hSBA titers were greater than or equal to (≥) 1:4 and ≥ 1:8. These analyses have been performed by the Health Protection Agency (HPA) laboratory.
Time Frame: At Month 69, one month post-booster vaccination
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 163 | 54
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 163 | 53
  hSBA-MenA, ≥ 1:4 | 163 | 46
  hSBA-MenC, ≥ 1:4: number analyzed (Participants) | 161 | 54
  hSBA-MenC, ≥ 1:4 | 161 | 54
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 156 | 52
  hSBA-MenW-135, ≥ 1:4 | 156 | 50
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 160 | 54
  hSBA-MenY, ≥ 1:4 | 160 | 52
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 163 | 53
  hSBA-MenA, ≥ 1:8 | 163 | 46
  hSBA-MenC, ≥ 1:8: number analyzed (Participants) | 161 | 54
  hSBA-MenC, ≥ 1:8 | 161 | 54
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 156 | 52
  hSBA-MenW-135, ≥ 1:8 | 156 | 50
  hSBA-MenY, ≥ 1:8 | 160 | 52

24. Secondary Outcome: Antibody Titers for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY
Description: as for outcome 9
Time Frame: At Month 69, one month post-booster vaccination
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 163 | 54
Titers
  hSBA-MenA: number analyzed (Participants) | 163 | 53
  hSBA-MenA | 1376.5 [1138.2 to 1664.6] | 101.2 [59.3 to 172.8]
  hSBA-MenC: number analyzed (Participants) | 161 | 54
  hSBA-MenC | 11986.8 [10085.2 to 14247.0] | 13692.2 [10094.2 to 18572.8]
  hSBA-MenW-135: number analyzed (Participants) | 156 | 52
  hSBA-MenW-135 | 14582.1 [12448.5 to 17081.5] | 235.7 [152.0 to 365.5]
  hSBA-MenY: number analyzed (Participants) | 160 | 54
  hSBA-MenY | 12835.9 [11074.4 to 14877.5] | 527.3 [356.5 to 779.9]

25. Secondary Outcome: Number of Subjects With a Vaccine Response to rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibodies
Description: Vaccine response to rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY was defined as rSBA antibody titers ≥1:32, for initially seronegative subjects (i.e. pre-vaccination rSBA antibody titers <1:8) and at least a 4-fold increase in rSBA antibody titers from pre to post-vaccination for initially seropositive subjects (i.e. pre-vaccination rSBA antibody titers ≥1:8).
Time Frame: At Month 69, one month post-booster vaccination
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 165 | 55
Participants
  rSBA-MenA | 147 | 54
  rSBA-MenC | 161 | 48
  rSBA-MenW-135 | 157 | 54
  rSBA-MenY | 156 | 54

26. Secondary Outcome: Number of Subjects With a Vaccine Response to hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibodies
Description: Vaccine response to hSBA-MenA, hSBA-MenC, rSBA-MenW-135 and hSBA-MenY was defined as hSBA antibody titers ≥ 1:8, for initially seronegative subjects (i.e. pre-vaccination hSBA antibody titers <1:4) and at least a 4-fold increase in hSBA antibody titers from pre to post-vaccination for initially seropositive subjects (i.e. pre-vaccination hSBA antibody titers ≥1:4).
Time Frame: At Month 69, one month post-booster vaccination
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 159 | 52
Participants
  hSBA-MenA | 156 | 43
  hSBA-MenC: number analyzed (Participants) | 156 | 50
  hSBA-MenC | 153 | 46
  hSBA-MenW-135: number analyzed (Participants) | 139 | 45
  hSBA-MenW-135 | 136 | 34
  hSBA-MenY: number analyzed (Participants) | 144 | 51
  hSBA-MenY | 142 | 35

27. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 50 millimeters (mm). "Any" was defined as incidence of the specified symptom regardless of intensity.
Time Frame: During the 4-day (Days 0-3) period following the booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in the primary 111414 study (NCT00674583) with the booster vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 171 | 60
Participants
  Any Pain | 113 | 35
  Grade 3 Pain | 7 | 4
  Any Redness | 62 | 25
  Grade 3 Redness | 8 | 4
  Any Swelling | 52 | 19
  Grade 3 Swelling | 4 | 3

28. Secondary Outcome: Number of Subjects With Any, Grade 3 and Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache and temperature (axillary temperature higher than [≥] 37.5 degrees Celsius [°C]). Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Fatigue = Fatigue that prevented normal activity. Grade 3 Gastrointestinal symptoms = Gastrointestinal symptoms that prevented normal everyday activities. Grade 3 Headache = Headache that prevented normal acitivity. Grade 3 Fever = Rectal temperature higher than (>) 39.5°C.
Time Frame: During the 4-day (Days 0-3) period following the booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in the primary 111414 study (NCT00674583) with the booster vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 169 | 58
Participants
  Any Fatigue | 38 | 12
  Grade 3 Fatigue | 3 | 0
  Related Fatigue | 28 | 10
  Any Gastrointestinal symptoms | 19 | 7
  Grade 3 Gastrointestinal symptoms | 2 | 1
  Related Gastrointestinal symptoms | 10 | 3
  Any Headache | 43 | 10
  Grade 3 Headache | 7 | 0
  Related Headache | 27 | 8
  Any Temperature | 11 | 5
  Grade 3 Temperature | 0 | 0
  Related Temperature | 9 | 3

29. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) period following the booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in the primary 111414 study (NCT00674583) with the booster vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 179 | 62
Participants | 26 | 8

30. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the 31-day (Days 0-30) period following the booster vaccination
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 179 | 62
Participants | 0 | 0

31. Secondary Outcome: Number of Subjects With Any New Onset of Chronic Illnesses (NOCIs)
Description: New onset of chronic illnesses (NOCIs) included: autoimmune disorders, asthma, type I diabetes and allergies.
Time Frame: During the 31-day (Days 0-30) period following the booster vaccination
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 179 | 62
Participants | 0 | 0

32. Secondary Outcome: Number of Subjects With Serious Adverse Events SAEs
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity.
Time Frame: Up to Month 32, 44, 56 and 68
Population: The analysis was performed on the Total Vaccinated cohort at Months 32, 44, 56 annd 68, which included all vaccinated subjects in the primary 111414 study (NCT00674583) who came back for persistence visit at Months 32, 44, 56 and 68, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Menjugate Group
Number analyzed (Participants) | 199 | 72
Participants
  Up to Month 32 | 0 | 0
  Up to Month 44: number analyzed (Participants) | 193 | 68
  Up to Month 44 | 0 | 0
  Up to Month 56: number analyzed (Participants) | 193 | 67
  Up to Month 56 | 0 | 0
  Up to Month 68: number analyzed (Participants) | 179 | 62
  Up to Month 68 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period; Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period; SAEs: during the entire study period (Month 32 up to Month 69).
Arm/Group | Nimenrix Group | Menjugate Group
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/179 | 0/62
Other Adverse Events (participants affected / at risk) | 130/179 | 48/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix Group (N=179) | Menjugate Group (N=62)
Erythema (Skin and subcutaneous tissue disorders) | 62 (62) | 25 (25)
Fatigue (General disorders) | 38 (38) | 12 (12)
Gastrointestinal disorder (Gastrointestinal disorders) | 19 (19) | 7 (7)
Headache (Nervous system disorders) | 43 (49) | 10 (10)
Pain (General disorders) | 113 (113) | 35 (35)
Pyrexia (General disorders) | 17 (17) | 8 (8)
Swelling (General disorders) | 52 (52) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.